CLINICAL TRIAL: NCT02510716
Title: Addressing Tobacco Use Disparities in Rural Older Adults Through an Innovative Mobile Phone Intervention: Testing the Feasibility of the Textto4gotobacco Intervention
Brief Title: Addressing Tobacco Use Disparities in Rural Older Adults Through an Innovative Mobile Phone Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Mayo Clinic (Other); Alliance for Clinical Trials in Oncology (Other); Duke Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00064813
Record Dates: First submitted 2015-07-24; First posted 2015-07-29 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-08

CONDITIONS: Tobacco Cessation
MeSH Terms: conditions — Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Scheduled Gradual Reduction (SGR) (Experimental): Four week SGR program plus support text messages.
  Interventions: Behavioral: SGR; Behavioral: Support message only
- Support Message Only (Active Comparator): Support text messages only.
  Interventions: Behavioral: Support message only

INTERVENTIONS:
Behavioral: SGR
  Arms: Scheduled Gradual Reduction (SGR)
Behavioral: Support message only

SUMMARY:
The purpose of this study is to evaluate the feasibility, acceptability and preliminary efficacy of a Scheduled Gradual Reduction (SGR) intervention via SMS (short message service) text messaging plus SMS Support Messages in decreasing smoking in an older adult rural population. The SGR group (n=20) will receive a four-week SGR program delivered via SMS text messages plus SMS support messages. The control group (n=20) will receive SMS support messages to aid in quitting.

ELIGIBILITY:
Inclusion Criteria:

1. Over 60 years of age,
2. Have smoked 100 cigarettes in their lifetime and currently smoke five or more cigarettes a day on average,
3. Have an address in a rural census tract defined by a RUCA code of 4-10,
4. Interested in participating in a cessation program,
5. Own a phone that has texting ability and free texting,
6. Have general knowledge of text messaging and
7. Are willing to receive and respond to text messages from the study teams, throughout the duration of the study.

Exclusion Criteria:

1. criteria include non-English speaking patients
2. already participating in a smoking cessation intervention study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Tobacco cessation, defined as quit rate at 30 days, as measured by self-reported abstinence from tobacco use | 30-days
  Quit rate at 30 days, as measured by self-reported abstinence from tobacco use

SECONDARY OUTCOMES:
Feasibility, as measured by proportion of return text messages | 30 days
  Proportion of return text messages sent per participants upon receiving "alert" text messages to use tobacco in the intervention group at 30 days Proportion of SMS support messages opened and/or read per participant
Acceptability, as measured by percentage of participants who reported that they would recommend the program to a friend | 30 days
  Percentage of participants who reported that they would recommend the program to a friend

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Noonan D, Silva S, Njuru J, Bishop T, Fish LJ, Simmons LA, Choi SH, Pollak KI. Feasibility of a text-based smoking cessation intervention in rural older adults. Health Educ Res. 2018 Feb 1;33(1):81-88. doi: 10.1093/her/cyx080. PMID 29309599